CLINICAL TRIAL: NCT02798731
Title: Physiologic Assessment of Microvascular Function and Its Impact on Cardiac Allograft Vasculopathy in Heart Transplant Patients: Prospective Registry and Pilot Study
Brief Title: Physiologic Assessment of Microvascular Function in Heart Transplant Patients
Status: Recruiting | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Joo Myung Lee, Assistant professor, Samsung Medical Center
Other Study IDs: HTPL2016-05-024
Record Dates: First submitted 2016-06-09; First posted 2016-06-14 (Estimated); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Cardiac Allograft Vasculopathy
Keywords: Heart transplant; Microvascular dysfunction; Cardiac allograft vasculopathy; Fractional flow reserve; Coronary flow reserve; Index of microvascular resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of the study is to evaluate the impact of early microvascular disease assessed by coronary physiologic indices such as fractional flow reserve (FFR), coronary flow reserve (CFR), index of microvascular resistance (IMR) on future occurrence of cardiac allograft vasculopathy (CAV) in heart transplant recipients.

DETAILED DESCRIPTION:
Cardiac allograft vasculopathy (CAV) or acute cellular rejection (ACR) are a leading cause of mortality and morbidity in heart transplant recipients. Most of the cases occur within 5 years after transplant and later incidence was known to be infrequent.

Mechanisms of CAV or ACR are thought to be multi-factorial involving both immunologic and non-immunologic factors that leads to injury of coronary endothelium and intimal hyperplasia. This unique mechanism results in long, diffuse and concentric stenosis of coronary arteries, different from those with conventional coronary atherosclerosis.

Due to lack of typical ischemic symptoms by denervated heart, diagnosis of CAV depends on routine screening tests rather than symptom based investigation. International Society for Heart and Lung Transplantation (ISHLT) guideline recommends annual or biannual coronary angiography screening until 5 years after transplant, but sensitivity of coronary angiography is limited because of diffuse involvement of all segments of coronary arteries. Alternatively, Intravascular ultrasound (IVUS) is a current standard for diagnosis and prognostication of CAV. It is well studied that progressive intimal thickening during the first year after transplant predicts future incidence of CAV and poor prognosis. However, the use of IVUS in the diagnosis of CAV is not generalized due to technical issues, high cost, procedure complications and ISHLT guideline states it is an option to exclude donor coronary artery disease, to detect rapidly progressive CAV, and provide prognostic information.

Recent development of single guidewire thermodilution technique enabled simple way to measure microvascular indices such as FFR, CFR, IMR. Our previous study shows, in patients with ischemic heart disease, presence of microvascular disease defined by low CFR and high IMR, predicts poor prognosis even without apparent epicardial disease. Considering its mechanism to involve diffuse coronary vasculature, CAV is believed to affect microvascular circulation in the early phase and spread to epicardial disease in its course. For this reason, by evaluating coronary physiology early after transplant, it may be possible to predict future progression of CAV.

There were previous studies which evaluated microvascular dysfunction in heart transplant patients. These studies indicated microvascular dysfunction at time of transplantation is related to progression of epicardial disease during first year after transplant, but lack of follow up prohibited from drawing any conclusion on occurrence of CAV later on. Another study by the same group evaluated microvascular dysfunction at 1 year after transplant and revealed it was associated with allograft vasculopathy at 5 years after transplant. However, this study did not evaluate impact of earlier assessments of microvascular dysfunction at time of transplantation on occurrence of CAV.

Therefore the current study will perform early physiologic assessments including fractional flow reserve, coronary flow reserve, and index of microcirculatory resistance in patients who received heart transplant and evaluate the impact of initial microvascular dysfunction on future occurrence of CAV or ACR during 6 years of follow up. The investigators hope to develop strong predictors of CAV or ACR that can be evaluated early after heart transplant and to improve outcome by preemptive therapy before overt development of the disease.

This study will be a pilot study and target sample size will be 200 consecutive patients to receive heart transplant.

ELIGIBILITY:
Inclusion Criteria:

* Subject over age of 18
* Patients received heart transplant

Exclusion Criteria:

* Patients with cardiogenic shock
* Patients with unstable vital sign that precludes coronary angiography
* Patients with major bleeding in last 3 months
* Patients with active bleeding
* Patients with coagulopathy
* Patients with severe valvular heart disease
* Patients who refused to provide informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients who received heart transplant undergoing coronary angiography for evaluation of coronary disease
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-05 (Actual); Primary Completion 2030-06 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Rates of cardiac death between patients with or without overt microvascular disease (CFR≤2 and IMR≥25) diagnosed with physiologic evaluation at 2-year follow-up after heart transplantation | 72 months
Acute cellular rejection between patients with or without overt microvascular disease | 72 months

SECONDARY OUTCOMES:
Occurrence of anatomically significant cardiac allograft vasculopathy (% diameter stenosis > 50% on CCTA) | 72 months
Comparison of total aggregated plaque volume and presence of adverse plaque characteristics on CCTA between transplant patients with or without overt microvascular disease (CFR≤2 and IMR≥25). | 72 months
Comparison of all-cause mortality in transplant patients with or without overt microvascular disease (CFR≤2 and IMR≥25) diagnosed with physiologic evaluation at 2-year follow-up after heart transplantation. | 24 months
Comparison of rates of cardiac death in transplant patients with or without overt microvascular disease (CFR≤2 and IMR≥25) diagnosed with physiologic evaluation at 1-year follow-up after heart transplantation. | 72 months
Comparison of IVUS and physiologic indices in prediction of CAV progression. | 72 months

CONTACTS AND LOCATIONS:
Overall Officials: Joo Myung Lee, MD, MPH, Principal Investigator — Samsung Medical Center; Jin-Oh Choi, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
After publication of first manuscript and trial results, the de-identified data will be shared by permission of principle investigator, when asked

REFERENCES:
- [Derived] Ha J, Lee SH, Choi KH, Shin D, Hong D, Kim D, Yang JH, Cho YH, Sung K, Park M, Kim JS, Park TK, Song YB, Hahn JY, Choi SH, Gwon HC, Oh JK, Choi JO, Lee JM. Microvascular Resistance Reserve and Prognosis After Heart Transplantation. JACC Cardiovasc Interv. 2025 Feb 24;18(4):439-452. doi: 10.1016/j.jcin.2024.11.011. PMID 40010915
- [Derived] Lee JM, Choi KH, Choi JO, Shin D, Park Y, Kim J, Lee SH, Kim D, Yang JH, Cho YH, Sung K, Choi JY, Park M, Kim JS, Park TK, Song YB, Hahn JY, Choi SH, Gwon HC, Oh JK, Jeon ES. Coronary Microcirculatory Dysfunction and Acute Cellular Rejection After Heart Transplantation. Circulation. 2021 Nov 2;144(18):1459-1472. doi: 10.1161/CIRCULATIONAHA.121.056158. Epub 2021 Sep 3. PMID 34474597
- [Derived] Lee SH, Choi KH, Lee JM, Hwang D, Rhee TM, Park J, Kim HK, Cho YK, Yoon HJ, Park J, Song YB, Hahn JY, Doh JH, Nam CW, Shin ES, Hur SH, Koo BK. Physiologic Characteristics and Clinical Outcomes of Patients With Discordance Between FFR and iFR. JACC Cardiovasc Interv. 2019 Oct 28;12(20):2018-2031. doi: 10.1016/j.jcin.2019.06.044. Epub 2019 Sep 25. PMID 31563683